CLINICAL TRIAL: NCT00297271
Title: Prospective Research in Memory Clinics (PRIME)
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CR004819; GALDEM4007 (Other: Janssen-Cilag Pty Ltd, Australia)
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Dementia; Mild Cognitive Impairment
Keywords: Dementia; Mild Cognitive Impairment; Patient Registries; Prospective Studies; Longitudinal Studies; Australia; Cholinesterase Inhibitors; Observational; Non-randomized
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mild cognitive impairment or dementia: Patients with mild cognitive impairment or dementia.
  Interventions: Other: Current treatment practice of each participating physician

INTERVENTIONS:
Other: Current treatment practice of each participating physician — Patients will be observed for the evaluation of current management strategies.

SUMMARY:
The purpose of the PRIME Study is to examine the current management and outcomes of patients with mild cognitive impairment or dementia. Approximately 4500 patients will be enrolled in this disease registry across 12 sites in Australia. Clinical, treatment, health status and economic data will be acquired over 3 years. The study will identify the relationships among demographic variables, prognostic features, geographic setting, treatment options and clinical, economic and health status (activities of daily living and caregiver impact) outcomes.

DETAILED DESCRIPTION:
A complete record of patient care will be collected to provide detailed information on the management and outcome of mild cognitive impairment and dementia and the profile of patients at participating sites. The data will be used to build models looking at the effect of management of these conditions on principal clinical events, health status and economic outcomes. This will provide the foundation for subsequent objective and prospective evaluation of evidence-based strategies for the optimal treatment of mild cognitive impairment and dementia in Australia. This study is not prescriptive, but will instead examine the influence of a whole range of routinely used management strategies on clinical and economic outcomes among mild cognitive impaired and dementia patients in Australia. This 'practice based' approach is increasingly widely used and is a useful tool for elucidating the relative effectiveness of different management strategies and for exploring relationships between patient characteristics, treatment and outcomes. Observational study - no study drug administered.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dementia under the DSM-IV criteria, or of Mild Cognitive Impairment, using the Peterson Criteria
* Living in the community (home, apartment or collective housing with nursing care available for less than 40 hours per week)
* Patient able to provide written informed consent, or provision of written informed consent by a legal guardian/proxy
* Availability of a caregiver willing to provide consent for required components of the study
* Fluent in English
* May be participating in a Phase IV or other post-marketing follow up study of an approved product for treatment of dementia

Exclusion Criteria:

* No concomitant life-threatening illness (a condition which is likely to interfere with the patient's ability to complete the study)
* Not unwilling or unable to complete the study
* Not concurrently participating in a clinical trial of an investigational drug (phase I, II or III)
* Unwillingness of patient or legal guardian / proxy to provide written informed consent
* Unwillingness of caregiver to provide written informed consent
* For patients with diagnosis of mild cognitive impairment: current or previous treatment with any cholinesterase or memantine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consenting patients with mild cognitrive impairement or dementia recruited at 12 participating sites accross Australia.
Sampling Method: Non-Probability Sample
Enrollment: 970 (Actual)
Dates: Start 2005-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to analyse the epidemiology and treatment outcomes of mild cognitive impairment and dementia under conditions of routine clinical practice | 6 months, 12 months and 36 months

SECONDARY OUTCOMES:
Change From Baseline in Clinical Dementia Rating Scale (total and overall score) | Baseline, 3, 6, 12, 24, and 36 months
  CDR is a 5-point scale to evaluates the clinical patterns and severity of the patients suspected or diagnosed as dementia in 6 areas: memory, orientation, judgment and problem solving ability, social activity, domestic living and hobbies, and hygiene and dressing up, where 0 = no cognitive impairment, 0.5 = very mild dementia, 1 = mild, 2 = moderate, and 3 = severe. Higher scores indicate worsening.
Mini Mental State Examination (total score) | Baseline, 3, 6, 12, 24 and 36 months
  The mini-mental state examination (MMSE) is a brief 30-point questionnaire test that is used or the assessment of dementia patients' cognitive impairment. Evaluation of points are as follows: 24 to 30 = no cognitive impairment, 18 to 23 = mild cognitive impairment, 0 to 17 = severe cognitive impairment. Lower scores indicate worsening.
The Alzheimer's Disease Assessment Scale (cognitive total score) | Baseline, 3, 6, 12, 24 and 36 months
  Alzheimer's Disease Assessment Scale is consists of 11 items, which assess memory, language and praxis, and can be administered independently of the non-cognitive portion. The total score ranges between 0 (best) and 70 (worst), with eight of the eleven items scoring between 0 (no impairment) and 5 (most impairment), and three of the items scoring from 0 to 8 (orientation questions), 0 to 10 (word recall) and 0 to 12 (word recognition). Higher scores indicate worsening
The Clock Drawing Test (total score) | Baseline, 3, 6, 12, 24 and 36 months
  The Clock Drawing Test is a simple and reliable measure of visuospatial ability. The test requires the participant to draw the face of a clock reading ten minutes after eleven, and the rater scores the result from 10 (best) to 1 (worst). Lower scores indicate worsening.
Frontal Assessment Battery (total score) | Baseline, 3, 6, 12, 24 and 36 months
  Frontal Assessment Battery is a short, simple testing for frontal lobe function that explores six domains of frontal lobe activity; conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental autonomy. It takes approximately 10 minutes to administer.
Functional Autonomy Measurement System (total score and subscores) | Baseline, 3, 6, 12, 24 and 36 months
  Functional Autonomy Measurement System is a 29-item scale developed according to the WHO classification of disabilities. It measures functional ability in five areas: activities of daily living (ADL), mobility, communication, mental functions and instrumental activities of daily living (IADL). For each item, the disability is scored on a 5-point scale: 0 (independent), -0.5 (with difficulty), -1 (needs supervision), -2 (needs help), -3 (dependent). A disability score (up to -87) can be calculated, together with sub-scores for each dimension.
Neuropsychiatric Inventory (total score, total distress to caregivers score, and total number of behaviors) | Baseline, 3, 6, 12, 24 and 36 months
  The neuropsychiatric inventory is used to characterize the neuropsychiatric symptom profiles in a variety of neurological diseases. Categories include symptoms like delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability, apathy, Night-time behaviour, appetite and eating, and aberrant motor activity. For each symptom, responder has to indicate "yes", if the symptom has been present since a month. The responder then rate the severity of the symptom on a 3-point scale for which scores range from "1 = Mild (noticeable, but not a significant change)" to "3 = Severe (very marked or prominent; a dramatic change)" and also rate the distress experienced due to the symptom on a 6-point scale for which scores range from "0 = Not distressing at all" to "5 = Extreme or very severe (extremely distressing, unable to cope with)". Higher scores indicate more behavioural disturbance.
Zarit caregiver burden interview (total score) | Baseline, 3, 6, 12, 24 and 36 months
  Zarit caregiver burden scale is used to measure caregiver burden as it relates to time, developmental comparison with peers, physical health, social relationships, and emotional health. It has 22 item and each question is scored on a 5-point Likert scale ranging from 0 = never present to 4 = nearly always present. The sum of the total scores of the 22-items is calculated in the range from 0 (low burden) to 88 (high burden). Higher scores indicate worsening.
Resource Utilization | Every month up to 36 months
  Resource utilization questionnaire will be completed at the end of each calendar month by participant/caregiver.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pty Ltd Clinical Trial, Study Director — Janssen-Cilag Pty Ltd
Locations (9):
- Australia (9):
  - Chermside
  - Fremantle
  - Geelong
  - Heidelberg
  - Hornsby
  - Kew
  - Newcastle
  - Randwick
  - Woodville

REFERENCES:
- See also: Prospective Research in Memory Clinics (PRIME) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=232&filename=CR004819_CSR.pdf